CLINICAL TRIAL: NCT01522898
Title: Cardiac Resynchronisation Therapy and AV Nodal Ablation Trial in Atrial Fibrillation
Brief Title: Cardiac Resynchronisation Therapy and AV Nodal Ablation Trial in Atrial Fibrillation Patients (CAAN-AF)
Acronym: CAAN-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Adelaide (Other)
Collaborators: Medtronic (Industry); Abbott Medical Devices (Industry); Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Prashanthan Sanders, Director, Centre for Heart Rhythm Disorders, University of Adelaide and Royal Adelaide Hospital, University of Adelaide
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAH-HREC-Protocol-#111234
Record Dates: First submitted 2012-01-25; First posted 2012-02-01 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Heart Failure; Atrial Fibrillation
Keywords: Heart Failure; Atrial Fibrillation
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medical Rate Control (Active Comparator): Medical Rate Control aimed at ventricular rate target of 90 beats per minute. Specific medical therapy to be determined for each patient by individual clinician.
  Interventions: Drug: Medical Ventricular Rate Control
- AV nodal ablation (Experimental): AV node ablation performed by percutaneous catheter ablation, with endpoint of complete heart block.
  Interventions: Procedure: AV nodal ablation

INTERVENTIONS:
Procedure: AV nodal ablation — Percutaneous catheter ablation of the AV node.
  Other Names: His Bundle Ablation, AV junctional ablation
  Arms: AV nodal ablation
Drug: Medical Ventricular Rate Control — Ventricular Rate Control with target ventricular rate of 90 beats per minute.
  Arms: Medical Rate Control

SUMMARY:
Cardiac resynchronization therapy (CRT) is a treatment for heart failure in patients who also suffer from ventricular dyssynchrony, a form of uncoordinated contraction of the ventricle (lower pumping chamber of the heart). In the past decade, CRT has become an established treatment for heart failure patients who are in normal rhythm, called sinus rhythm. An important subset of heart failure patients are those with atrial fibrillation (AF), who make up around 1 in 4 HF patients, and are over-represented amongst HF patients with more advanced symptoms. In heart failure patients with AF, CRT has proven not to be as effective as in sinus rhythm, due to competition between beats generated by the CRT device and beats conducted from the heart's own electrical conduction system. In the current study, we aim to test the hypothesis that ablating the AV node, which controls electrical conduction from the heart's atria (top chamber) to its ventricles (lower chambers), will improve survival and heart failure symptoms in CRT patients with co-existent AF. The results are important, because they will provide a way of passing on the benefits of CRT, such as improved survival, less heart failure symptoms, and better quality of life, to heart failure patients who also suffer from AF.

DETAILED DESCRIPTION:
Background: Cardiac Resynchronization Therapy (CRT) is an established treatment in heart failure (HF) patients with ventricular dyssynchrony who remain in sinus rhythm. Available clinical data has shown inferior outcomes of CRT in HF patients with co-existent atrial fibrillation (AF), who comprise up to 27% of HF patients, and are over-represented in advanced HF classes. We hypothesize, based on the results of a systematic review we recently published in the Journal of the American College of Cardiology, that AV nodal ablation may improve survival, heart failure and functional outcomes in CRT recipients with co-existent AF.

Design: This study will be a multicentre, prospective, randomized controlled trial. Patients with ischemic or nonischemic cardiomyopathy heart failure (NYHA II, III or ambulatory class IV), left ventricular dysfunction (EF ≤ 35%), prolonged intraventricular conduction (QRS duration ≥ 120ms), and persistent or permanent AF will be considered for the study. Persistent AF will be defined as patients where obtaining and maintaining sinus rhythm is deemed either not worthwhile, or to be ineffective in the long term, or where both the patient and the physician accept the presence of AF, where rhythm control intervention is, by definition, no longer pursued. Permanent AF is defined as AF where sinus rhythm cannot be restored.

Eligible subjects will be randomized into one of two arms: (1) CRT-D plus AV nodal ablation ("AV nodal ablation arm [AVNA]") or (2) CRT-D alone ("rate control arm").

Enrollment: 590 subjects, with 295 subjects in the AV node ablation arm and 295 subjects in the control arm, will be enrolled. Study patients will undergo stratified randomization at ≥ 30 days after CRT implant. Participants in will sign informed consent and be screened prior to randomisation. After CRT implant, patients will have at least 30 days for optimisation of heart failure therapy, prior to randomisation.

Randomisation: A computer-generated web-based randomisation schedule will be used. Randomisation will be stratified by trial centre. Randomisation is considered the trial entry point.

Outcomes: The primary endpoint is a composite of all cause mortality and non-fatal heart failure events. Secondary endpoints include all-cause mortality, cardiovascular mortality (including classification in terms of suddenness and arrhythmic mechanism by prespecified Hinkle-Thaler criteria), non-fatal heart failure events, 6-minute walking test distance, quality of life, unplanned hospitalization, and ventricular arrhythmias requiring device therapy, inappropriate shocks, cardiovascular MRI prediction of response, percentage pacing and prediction of response to therapy, ventricular reverse remodeling.

Statistical Plan: The study is powered to find a 25% relative reduction in event rate, with sample sizes calculated assuming a two-tailed α=0.05,1-β=0.80, and 10% sample size increment allow for to drop in the event rate (AV nodal ablation arm), drop out or cross-over (feasibly, control to AVNA arm only). It is planned to perform three interim (0.25, 0.5 0.75 information fractions) and a final analysis requiring 295 patients per arm with a final P-value at ≤ 0.045; stopping rules according to the method of O'Brien and Fleming. The boundaries (z scores: ±4.332, ±2.963, ±2.359, ±2.014; and nominal P-values: 0.000015, 0.0031, 0.014, 0.044)) were derived using the statistical package PASS (V12). Outside of these defined analyses, the Data Safety Monitoring Board (DSMB) will have access to data reports and will be able to stop the trial at any time.

All analyses will be based on the intention-to-treat principle. The primary (binary) mortality-outcome will be analysed using the Cochran-Mantel-Haenszel statistic and logistic regression with pre-specified (baseline) covariates. Time-to-event analyses will be initially undertaken by the Kaplan-Meier survival analysis approach. Key secondary outcomes such as all-cause mortality, cardiovascular mortality, unplanned hospitalisation, and rates of ventricular arrhythmia episodes will be analysed using either Cox proportional hazards models or Fine and Gray competing risks regression as appropriate. Continuous secondary outcomes such as the 6-minute walking distance, Short Form 36 (SF36) scores, Minnesota Living with Heart Failure (MLWHF) score will be compared between randomised groups over time using linear mixed effects models.

Significance and Impact: The study will answer a central clinical question directly impacting the care of HF patients with AF, and will be expected to change current HF management guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Persistent (≥ 1 month) or permanent atrial fibrillation. Persistent AF will be where obtaining and maintaining sinus rhythm is deemed either not worthwhile, or to be ineffective in the long term, or where both the patient and physician accept the presence of AF, where rhythm control intervention is, by definition no longer pursued. Permanent AF is defined as atrial fibrillation where sinus rhythm cannot be restored.
* NYHA class II , III or ambulatory class IV heart failure
* Left Ventricular Ejection Fraction (LVEF) ≤ 35% by objective criteria such as echocardiography, or cardiac MRI
* QRS duration on 12-lead ECG ≥ 120ms
* Able and willing to comply with all pre-, post- and follow-up testing and requirements.

Exclusion Criteria:

* age < 18 years
* pregnancy
* previous AV nodal ablation
* Second or third degree AV block
* Inability to provide informed consent
* life expectancy less than 24 months due to co-morbid illness other than heart failure erg cancer, end-stage renal disease, liver failure
* Paroxysmal Atrial Fibrillation that self terminates within 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2013-03; Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
All-cause mortality and non-fatal heart failure events | Final-analysis at completion of recruitment and follow-up period (minimum 2 year follow-up)
  This is a composite of all-cause mortality and non-fatal heart failure events. All-cause mortality will be determined by a designated clinical events committee.
  Heart Failure events will be documented by clinical data from the hospital In CAAN-AF, a subject will be described as having a "Heart Failure Event" when the subject has symptoms and/or signs consistent with congestive heart failure and:
  * responsive to parenteral diuretic or inotropic support as an outpatient
  * responsive to oral or parenteral diuretic or inotropic support during an inpatient stay

SECONDARY OUTCOMES:
All-cause mortality | Final-analysis at completion of recruitment and follow-up period (minimum 2 year follow-up)f recruitment
  All-cause mortality will be determined after adjudication committee review of clinical records, and death certificate data.
Cardiovascular mortality | Final-analysis at completion of recruitment and follow-up period (minimum 2 year follow-up)
  Cardiovascular deaths will be classified in terms of suddenness and arrhythmic mechanism according to the Hinkle-Thaler criteria.
Non-Fatal Heart Failure Events | Final-analysis at completion of recruitment and follow-up period (minimum 2 year follow-up)
  Heart Failure events will be documented by clinical data from the hospital In CAAN-AF, a subject will be described as having a "Heart Failure Event" when the subject has symptoms and/or signs consistent with congestive heart failure and:
  * responsive to parenteral diuretic or inotropic support as an outpatient
  * responsive to oral or parenteral diuretic or inotropic support during an inpatient stay
6-minute walking distance | Final-analysis at completion of recruitment and follow-up period (minimum 2 year follow-up)
  6-minute walking distance will be measured according to standard criteria.
Quality of Life questionnaires | Final-analysis at completion of recruitment and follow-up period (minimum 2 year follow-up)
  Quality of life as assessed by the Short Form 36 (SF-36) questionnaire and Minnesota Living with Heart Failure Questionnaire
Unplanned Hospitalization | Final-analysis at completion of recruitment and follow-up period (minimum 2 year follow-up)
  Unplanned hospital admissions will be assessed by a combination of patient self-report, hospital record and/or treating physician interrogation. The reason, date and duration of hospitalization will be recorded Planned hospitalizations (hospital visits for elective or planned medical interventions) will excluded from this outcome
Ventricular arrhythmias requiring device therapy | Final-analysis at completion of recruitment and follow-up period (minimum 2 year follow-up)
  Ventricular arrhythmias requiring device therapy will be determined by implantable Cardioverter Defibrillator (ICD) interrogation records and clinical records. At each site, the number, duration and type (VT/VF) of device recorded arrhythmias will be recorded, as well as the need for device therapy (anti-tachycardia pacing and/or ICD shocks).

OTHER OUTCOMES:
Inappropriate shocks | Final-analysis at completion of recruitment and follow-up period (minimum 2 year follow-up)
  The clinical events committee will review clinical records to ascertain if device therapies are appropriate or inappropriate.
Cardiovascular MRI prediction of response | Final-analysis at completion of recruitment and follow-up period (minimum 2 year follow-up)
  Cardiovascular MRI will be performed in subjects eligible for this procedure prior to implantation of CRT device, when available. Cardiovascular MRI data will be evaluated for the ability to predict clinical CRT response.
Depression | Final-analysis at completion of recruitment and follow-up period (minimum 2 year follow-up)
  Depression will be evaluated in all patients at specified clinical follow-up visits with the Center for Epidemiologic Studies Depression Scale (CES-D questionnaire).
Ventricular reverse remodelling | Final-analysis at completion of recruitment and follow-up period (minimum 2 year follow-up)
  Left ventricular reverse remodeling will be assessed by echocardiographic parameters including left ventricular end systolic volume, left ventricular ejection fraction. An echocardiography core laboratory has been established to process images from individual trial sites for this purpose.

CONTACTS AND LOCATIONS:
Overall Officials: Prashanthan Sanders, MBBS PhD, Principal Investigator — University of Adelaide
Locations (33):
- Australia (23):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - Concord Hospital, Concord, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Fiona Stanley, Murdoch, Perth, WA
  - Royal Brisbane Hospital, Brisbane, Queensland
  - Prince Charles Hospital, Chermside, Queensland
  - Townsville Hospital and Health Service, Douglas, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Monash Medical Centre, Clayton, Victoria
  - Geelong Hospital, Geelong, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Melbourne Private Hospital, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Sir Charles Gairdner Hospital, Perth, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Germany (4):
  - Universitätsmedizin Mainz, Mainz, Gebäude 401/k
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg, Martinistr. 52 Gebäude Ost 50, 8. OG, Raum 842
  - University Clinic of Cologne, Cologne
  - Asklepios Hospital, St. Georg
- National Heart Institute, Kuala Lumpur, Malaysia
- New Zealand (4):
  - Tauranga Hospital, Tauranga, Bay of Plenty
  - Auckland City Hospital, Auckland
  - Waikato Hospital, Hamilton
  - Wellington Hospital, Wellington
- James Cook University Hospital, Middlesbrough, United Kingdom